CLINICAL TRIAL: NCT03317015
Title: A Randomized, Double-blind, Parallel-group, Multicenter, Phase III Prospective Non-inferiority Clinical Trial to Assess Efficacy and Safety of Nasacort® Nasal Spray (Triamcinolone, 55µg) in Comparison With Flixonase® Nasal Spray (Fluticasone, 50 µg) in Adults Suffering From PAR (Perennial Allergic Rhinitis) Administered Once a Day for 28 Days
Brief Title: A Study to Assess Efficacy and Safety of Nasacort® Nasal Spray in Comparison With Flixonase® Nasal Spray in Adults Suffering From Perennial Allergic Rhinitis (PAR)
Acronym: NASANIF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRICAL07830; U1111-1178-4882 (Other: UTN)
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Rhinitis Allergic
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Triamcinolone; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Nasacort® (Experimental): Nasacort® will be sprayed twice in each nostril once every morning
  Interventions: Drug: triamcinolone XRG5029
- Group B - Flixonase® (Active Comparator): Flixonase® will be sprayed twice in each nostril once every morning
  Interventions: Drug: fluticasone

INTERVENTIONS:
Drug: triamcinolone XRG5029 — Pharmaceutical form: spray solution
  Route of administration: nasal
  Other Names: Nasacort®
  Arms: Group A - Nasacort®
Drug: fluticasone — Pharmaceutical form: spray solution
  Route of administration: nasal
  Other Names: Flixonase®
  Arms: Group B - Flixonase®

SUMMARY:
Primary Objective:

* To assess efficacy of Nasacort® (triamcinolone) nasal spray, 55 µg per dose, in comparison with Flixonase® (fluticasone) nasal spray, 50 µg per dose, by reflective total nasal symptom score (rTNSS) (24 h) after 28 days of treatment compared with baseline (0 day of treatment) in adult patients suffering from PAR (perennial allergic rhinitis).

Secondary Objectives:

* To evaluate safety of Nasacort® (triamcinolone) nasal spray, in comparison with Flixonase® (fluticasone) administered for 28 days by assessment of adverse events reports.
* To evaluate patient and physician satisfaction after 28 days of treatment by 5-point scale.
* To estimate improvement of quality of life during the study by mini Rhinoconjunctivitis Quality of Life Questionnaire (miniRQLQ).

DETAILED DESCRIPTION:
The total study duration per patient will be up to approximately 33 days.

ELIGIBILITY:
Inclusion criteria:

* Females and males ≥18 and ≤50 years old.
* Patients with previously diagnosed PAR with a positive skin prick test response to an appropriate allergen performed not earlier than 12 months prior to the Screening visit.
* Patients must be clinically symptomatic (rTNSS reflecting symptoms for the previous 24 h ≥8 with two or more symptoms rated as moderate or severe).
* Negative urine pregnancy test during screening before first dose of study medication is administered in women with child-bearing potential.
* Women must use an effective contraceptive method during the study period.
* Patients should be able to understand the study, including risks and adverse events; collaborating with Investigator and proceed according with protocol.
* Signed informed consent form.

Exclusion criteria:

* Compromised ability to provide informed consent.
* Participation in any other clinical study.
* History of severe local reaction(s) or anaphylaxis to skin testing.
* Upper respiratory tract or sinus infection that required antibiotic therapy without at least a 14-day washout prior to the Screening Visit, or viral upper respiratory infection within 2 weeks prior to the Screening Visit.
* Subjects who have used any drug (Flixonase or Nasacort) in an investigational protocol 4 weeks prior to the Screening Visit.
* Female subjects who are breast-feeding, pregnant, or intend to become pregnant.
* Patients with nasal abnormalities, including nasal polyps, and marked septum deviation that interferes with nasal airflow.
* Recent (in the last 3 months) or unhealed nasal septum ulcers, nasal surgery, or nasal trauma.
* Specific immunotherapy finished later than 6 months prior to Visit 1.
* Use of following medications:

  * Intranasal corticosteroids within 4 weeks prior to Visit 1;
  * Inhaled, oral, intramuscular, intravenous, ocular, and/or dermatological corticosteroid within 8 weeks prior to Visit 1;
  * Cromones within 2 weeks prior to Visit 1;
  * Short-acting antihistamines, including antihistamines contained in insomnia formulations within 3 days prior to Visit 1;
  * Long-acting antihistamines within 10 days prior to Visit 1: loratadine, desloratadine, fexofenadine, cetirizine;
  * Intranasal antihistamines within 2 weeks prior to Visit 1;
  * Intranasal, oral, or inhaled anticholinergics within 3 days prior to Visit 1;
  * Oral antileukotrienes within 3 days prior to Visit 1;
  * Use of immunosuppressive medications 8 weeks prior to screening.
* Patients allergic to or have sensitivity to the study drug (triamcinolone acetonide, fluticasone propionate) or its excipients.
* Patients suffering from SAR (seasonal allergic rhinitis).
* Patients suffering from non-allergic rhinitis.
* Patients suffering from rhinitis medicamentosa.
* Patients suffering from non-allergic rhinitis caused by viral, bacterial etc infection.
* Patients suffering from bronchial asthma.
* Patients suffering from chronic sinusitis.
* In case of non-allergic rhinitis, nasal trauma or other condition that during the study can interfere with symptoms evaluation, subject would be excluded from the study.
* Patients with physical impairment that would affect subject's ability to participate safely and fully in the study.
* Clinical evidence of a Candida infection of the nose.
* History of psychiatric disease, intellectual deficiency, poor motivation, substance abuse (including drug and alcohol) or other conditions that will limit the validity of informed consent or that would affect the proper daily diary filling.
* Previous history and/or current diagnosis of glaucoma and cataract.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total nasal symptom score | From baseline (0 day of treatment) to 28th day of treatment

SECONDARY OUTCOMES:
Change from baseline in quality of life questionnaire scores (miniRQLQ questionnaire) | From baseline (0 day of treatment) to 28th day of treatment
Number of participants with adverse events | From baseline (0 day of treatment) to 28th day of treatment
Assessment of patient satisfaction using the 5-point scale questionnaire | 28th day of treatment
Assessment of physician satisfaction using the 5-point scale questionnaire | 28th day of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org